CLINICAL TRIAL: NCT00253929
Title: The Influence of the 1976T>C Polymorphism in the Adenosine A2A Receptor Gene on Adenosine-Induced Vasodilation and the Influence of the 34C>T Polymorphism in the AMP Deaminase Gene on Post-Occlusive Reactive Hyperemia.
Brief Title: Effect of Polymorphisms in the Adenosine a2a Receptor Gene and AMPD2 Gene on Adenosine-Induced Vasodilation and Reactive Hyperemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SNPAdenosine; ZonMw Nr. 920-03-249
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2006-02

CONDITIONS: Blood Flow in Healthy Volunteers
Keywords: adenosine; polymorphisms; blood flow; adenosine A2a receptor; AMP deaminase

INTERVENTIONS:
Drug: Intra-arterial infusion of adenosine
Drug: intra-arterial infusion of caffeine
Drug: intra-arterial infusion of acetylcholine
Drug: intra-arterial infusion of sodium nitroprusside
Procedure: Occlusion of arm-circulation by inflation of upper-arm cuff to 200mmHg for 2, 5 and 13 minutes

SUMMARY:
The endogenous nucleoside adenosine can induce various cardiovascular and neurohumoral effects by stimulation of specific adenosine receptors. taken together these effects protect against ischaemia-reperfusion injury of (myocardial)muscles and agsinst the development of atherosclerosis. Genetic variations in genes encoding for adenosine receptors or for enzymes involved in the formation or breakdown of adenosine could potentially modulate these effects. In this study, we aim to determine the functional effects of two frequent genetic polymorphisms in the adenosine receptor and AMPdeaminase (involved in the formation of adenosine) on the vascular effects of adenosine.

DETAILED DESCRIPTION:
The endogenous nucleoside adenosine can induce various cardiovascular and neurohumoral effects by stimulation of specific adenosine receptors. taken together these effects protect against ischaemia-reperfusion injury of (myocardial)muscles and agsinst the development of atherosclerosis. Genetic variations in genes encoding for adenosine receptors or for enzymes involved in the formation or breakdown of adenosine could potentially modulate these effects. In this study, we aim to determine the functional effects of two frequent genetic polymorphisms in the adenosine receptor and AMPdeaminase (involved in the formation of adenosine) on the vascular effects of adenosine.

In 100 healthy young volunteers, we will determine the genotype of the adenosine A2A receptor gene. We expect to find approximately 15 subjects with the 1976T>C polymorphisms. It is known that this polymorphism is associated with an increased neuropsychological sensitivity to caffeine administration.

We will explore whether this polymorphism is associated with a different vasodilating response to the administration of adenosine and caffeine into the brachial artery. Blood flow will be measured with venous occlucion plethysmography.

Secondly, we will also determine the genotype of the AMPD1 gene. We expect to find 15 subjects with the 34C>T mutation, which is a loss-of-function-mutation. Cardiovascular patients with this mutation are known to have a survival benefit. We will explore whether the post-occlusive reactive hyperemia in the forearm is potentiated, because during ischaemia, more adenosine is formed in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 year

Exclusion Criteria:

* hypertension
* diabetes
* cardiovascular or pulmonary disease
* asthma

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2005-11; Study Completion 2006-02

PRIMARY OUTCOMES:
A2A: adenosine- and caffeine induced vasomotion (blood flow)
AMPD:post-occlusive reactibe hyperemic blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Principal Investigator — Radboud University Medical Center; Paul Smits, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Riksen NP, Franke B, van den Broek P, Naber M, Smits P, Rongen GA. The 22G>A polymorphism in the adenosine deaminase gene impairs catalytic function but does not affect reactive hyperaemia in humans in vivo. Pharmacogenet Genomics. 2008 Oct;18(10):843-6. doi: 10.1097/FPC.0b013e328305e630. PMID 18794722